CLINICAL TRIAL: NCT01746446
Title: LifeCourse: A Supportive Care Approach for Patients Late in Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Collaborators: Robina Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38632
Record Dates: First submitted 2012-11-27; First posted 2012-12-11 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Ongoing or Significant Medical Condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care team (Experimental): Patients are offered the support and services of the care team.
  Interventions: Other: Care team
- Usual Care (No Intervention): Patients receive usual care.

INTERVENTIONS:
Other: Care team — Provides additional support to patients, family, and friends.
  Arms: Care team

SUMMARY:
The purpose of the study is to test a new model of care for patients with an ongoing or significant medical condition.

DETAILED DESCRIPTION:
LifeCourse is a late life care approach that promotes whole person care through a structured approach built upon an expanded set of palliative care domains and chronic illness care practices. It includes a trained lay healthcare worker as the primary contact who follows the patient across care settings and over time. The care guide asks patients and caregivers to articulate individualized goals and take part in decision making, and uses a family-oriented approach to understand needs, leverage strengths, and empower families to effectively support the individual living with serious illness.

ELIGIBILITY:
Inclusion criteria

* Patient has an Allina Health primary or specialty provider
* Patient's medical chart indicates an on-going or significant medical condition
* LifeCourse will invite vulnerable patients to enroll, including:
* Critically ill patients
* Cognitively impaired patients
* Elderly patients, some of whom may have cognitive impairment and/or be institutionalized

Exclusion Criteria

* Patient resides in a zip code which does not lie partially within a 45 mile radius from the Allina Health Commons in Minneapolis, Minnesota.
* Patient has not visited an Allina facility, affiliate, or community partner within the last year.
* Patient is eligible for hospice.
* Patient is actively dying.
* Patient is abusive or is discharged against medical advice (AMA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Patient Quality of Life | Change from baseline survey responses at 3 month intervals until subject withdrawal or date of death from any cause, whichever comes first, up to six years.
  Patient QOL was measured using the Functional Assessment of Chronic Illness Therapy-Palliative v4 (FACIT-Pal) survey, a general measure of health-related QOL in 4 domains: physical, social, emotional, and functional, plus a measure of end-of-life experiences. Items were reverse scored according to scoring guidelines and domain scores were calculated via prorated scores when there were <50% missing items for a given domain and <20% missing domains for a total score.
Patient Care Experience | Change from baseline survey responses at 3 month intervals until subject withdrawal or date of death from any cause, whichever comes first, up to six years.
  Patient care experience was collected via a previously validated survey tool focused on the patient's experience with their care team in the last 30 days. Three domains were scored: care team, goals, and communication with prorated scores when there were <50% missing items for a given domain and <20% missing domains for a total score.
Caregiver care experience | Change from baseline survey responses at 3 month intervals until subject withdrawal or date of death from any cause, whichever comes first, up to six years.
  Caregiver care experience was measured by a developed tool, addressing various aspects of care experience. An overall score was calculated by summing answers to all items. Scores were also calculated in 3 domains: care team, communication, and support.
Caregiver Quality of Life | Change from baseline survey responses at 3 month intervals until subject withdrawal or date of death from any cause, whichever comes first, up to six years.
  aregiver QOL was assessed via the patient-reported outcomes measurement information system (PROMIS) which asks caregivers to report their QOL in 8 domains. The PROMIS-29 scores were calculated by summing answers to all items within each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Eric W Anderson, MD, Principal Investigator — Allina Health
Locations (3):
- United States (3):
  - Augustana Health Care Center, Minneapolis, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Walker Methodist Health Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schellinger S, Cain CL, Shibrowski K, Elumba D, Rosenberg E. Building New Teams for Late Life Care: Lessons From LifeCourse. Am J Hosp Palliat Care. 2016 Jul;33(6):561-7. doi: 10.1177/1049909115574692. Epub 2015 Mar 5. PMID 25747670
- [Background] Fernstrom KM, Shippee ND, Jones AL, Britt HR. Development and validation of a new patient experience tool in patients with serious illness. BMC Palliat Care. 2016 Dec 30;15(1):99. doi: 10.1186/s12904-016-0172-x. PMID 28038669
- [Background] Anderson EW, Frazer MS, Schellinger SE. Expanding the Palliative Care Domains to Meet the Needs of a Community-Based Supportive Care Model. Am J Hosp Palliat Care. 2018 Feb;35(2):258-265. doi: 10.1177/1049909117705061. Epub 2017 Apr 20. PMID 28423918
- [Background] Anderson EW, White KM. "It Has Changed My Life": An Exploration of Caregiver Experiences in Serious Illness. Am J Hosp Palliat Care. 2018 Feb;35(2):266-274. doi: 10.1177/1049909117701895. Epub 2017 Apr 16. PMID 28413927
- [Background] Schellinger SE, Anderson EW, Frazer MS, Cain CL. Patient Self-Defined Goals: Essentials of Person-Centered Care for Serious Illness. Am J Hosp Palliat Care. 2018 Jan;35(1):159-165. doi: 10.1177/1049909117699600. Epub 2017 Mar 23. PMID 28330379
- [Background] Shippee ND, Shippee TP, Mobley PD, Fernstrom KM, Britt HR. Effect of a Whole-Person Model of Care on Patient Experience in Patients With Complex Chronic Illness in Late Life. Am J Hosp Palliat Care. 2018 Jan;35(1):104-109. doi: 10.1177/1049909117690710. Epub 2017 Jan 29. PMID 28133973
- [Background] Cain CL, Taborda-Whitt C, Frazer M, Schellinger S, White KM, Kaasovic J, Nelson B, Chant A. A mixed methods study of emotional exhaustion: Energizing and depleting work within an innovative healthcare team. J Interprof Care. 2017 Nov;31(6):714-724. doi: 10.1080/13561820.2017.1356809. Epub 2017 Sep 18. PMID 28922038
- [Background] Anderson EW, White KM. "This Is What Family Does": The Family Experience of Caring for Serious Illness. Am J Hosp Palliat Care. 2018 Feb;35(2):348-354. doi: 10.1177/1049909117709251. Epub 2017 Jun 30. PMID 28662594
- [Derived] Britt HR, JaKa MM, Fernstrom KM, Bingham PE, Betzner AE, Taghon JR, Shippee ND, Shippee TP, Schellinger SE, Anderson EW. Quasi-Experimental Evaluation of LifeCourse on Utilization and Patient and Caregiver Quality of Life and Experience. Am J Hosp Palliat Care. 2019 May;36(5):408-416. doi: 10.1177/1049909118817740. Epub 2018 Dec 13. PMID 30541333

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT01746446/Prot_SAP_000.pdf
  • Informed Consent Form (2014-09-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT01746446/ICF_001.pdf